CLINICAL TRIAL: NCT04923854
Title: Phenotypic Exploration of Autism Spectrum Disorders Retrospective and Prospective Data
Acronym: EXPECT
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP191023
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2021-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Autism Spectrum Disorders (ASD) are a heterogeneous group of severe developmental abnormalities of the nervous system characterized by deficits in social interaction and verbal and nonverbal communication affecting approximately 1% of the general population.

In 5-40% of cases, genetic factors are identified as the cause of these disorders.

Despite this unique definition and the advancement of techniques, ASD is still a clinically and genetically heterogeneous condition, as several hundred genes have been identified to date.

Primary Objective and Endpoint Primary Objective:

Exploration of phenotypic heterogeneity in patients with ASD.

Primary endpoint:

* Routine Care Clinical Investigation Criteria.
* Scores on assessment scales,

DETAILED DESCRIPTION:
Autism Spectrum Disorders (ASD) are a heterogeneous and severe developmental abnormalities of the nervous system characterized by deficits affecting social interactions and verbal and nonverbal communication (DSM-5, 2013), affecting approximately 1% of the general population (Brugha, 2012). In 5-40% of cases, genetic factors are identified as the cause of these disorders, prevalence depending on the technique used (Exome and/or SNPs Array) and the associated intellectual deficit. In the majority of cases, the etiology remains unknown. The familial aggregation of ASDs and the significant excess of concordant monozygotic twins over dizygotic twins demonstrate the strong involvement of genetic factors in autism. Studies of microdeletions/microduplications (copy number variants) or by Whole Exome Sequencing and Whole Genome Sequencing (Single Nucleotide Variants) show the involvement of many genes in the predisposition to autism. However, ASD remains a clinically and genetically heterogeneous disorder, since several hundred genes have been identified to date.

The main objective of our project is to allow the retrospective and prospective collection of data on the phenotypic and genetic characterization of ASD patients in a structured way in order to allow the development of a new dynamic in terms of research. The identification of genetic factors (Delorme et al, Nature Medicine, 2013) and biological pathways involved in the emergence of autistic symptoms (Bourgeron, Nature Neuroscience 2015) is fundamental. The identification of biological pathways is an indispensable step for the development of new therapeutic strategies. In addition, a major challenge of this study is to better understand the phenotype/genotype relationships in ASD. This requires the constitution of a large cohort of patients taking into account their multimodal, extensive and precise exploration of clinical, neuroanatomical (MRI, EEG) and biological phenotypes and to correlate them with genetic data.

The work carried out by our teams and collaborators has led to the identification of numerous genes associated with ASD and involved in synaptic formation and regulation: NLGN3-4 (Jamain et al, Nature Genetics 2003), SHANK1-3 (Durand el al Nature Genetics 2007, Sato et al Am J Hum Genet 2013, Leblond et al Plos Genetics 2013, 2014), CNTN-6 (Mercati et al Mol Psychiatry 2016) and CNTNAP4 (Karayannis, Nature, 2014) (for review Toro et al, TIGS 2012; Delorme et al, Nature Medicine ,2013; Bourgeron, Nature Neuroscience 2015). This work was combined with extensive phenotypic explorations of patients and their relatives. It has allowed us to specify the neuroanatomical characteristics of the patients (Lefebvre et al. Biol Psychiatry 2014) and their genetic substrate (Toro et al, Mol Psychiatry 2015), but also the underlying cognitive processes (Dumas et al, PNAS, 2014; Zalla et al. Cortex 2014, 2015; Grezes et al Hum Brain Mapp, 2014). More recently, we have shown the existence of abnormalities in the regulation of the melatonin synthesis pathway (Pagan et al, TransPsychiatry 2014; Pagan et al, J pineal Res 2015) or immunological abnormalities (in particular HLA anomalies (Bennabi et al, 2018)

Description of the population to be studied and rationale for its choice

We wish to explore the heterogeneity of autism spectrum disorders in a population received in routine care in our evaluation units. These are patients followed in the Child and Adolescent Psychiatry Department at the Robert Debré Hospital in Paris, who meet the diagnostic criteria of ASD according to DSM-5, aged 0 to 17 years.

Description of the element(s) on which the research focuses

The main objective of our project is to explore the phenotypic heterogeneity of ASD. The collection of data from the routine clinical evaluation of a large number of subjects will allow for a better phenotypic and genetic characterization of patients in a structured manner to allow for the development of a new dynamic in terms of research. We wish to carry out a non-interventional, mono-centric study based on data from the evaluation of patients in clinical practice.

To allow this work we must favour:

1. the collection of phenotypic data of the patients evaluated in our service, including

   * Clinical phenotypes: standardized evaluation of phenotypes in clinical practice, according to current recommendations
   * Neuroanatomical phenotypes: brain imaging (MRI), electrophysiology EEG, Eye-Tracking,
   * Biological phenotypes: serological, genetic of patients hospitalized in our department;
2. the linking of these data via a database regrouping this information (or allowing them to be grouped);
3. the development of a new dynamic in terms of translational research concerning ASD.

The creation of this cohort, based on data from the evaluation done in clinical practice, will help identify biological pathways involved in autism, the development of new therapeutic strategies for patients and a more personalized medicine.

Justification of the duration of the research.

The total duration of the research will be 6 years (5 years of inclusion and a maximum of 12 months of patient observation), renewable by possible extension of the study.

This duration will allow the collection of data from the evaluation of approximately 300 patients per year (i.e. 1500 patients over the next 5 years). This study duration is essential to collect a sufficient number of patients to have enough statistical power for the study. Also the extensive phenotypic and genetic exploration requires - in order to be able to cross-reference the data and establish relevant subgroups - to have large samples of subjects.

ELIGIBILITY:
Inclusion Criteria:

* child (age <18 years) with Autism Spectrum DisorderAutism Spectrum Disorder

Exclusion Criteria:

-

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: child (age <18 years) with Autism Spectrum Disorder
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
The main objective is to better understand the phenotypic heterogeneity of Autism Spectrum Disorder (ASD). | 12 months
  DSM5 (Diagnostic statistical Manual of Mental disorders) Autism diagnostic scales

CONTACTS AND LOCATIONS:
Overall Officials: Richard DELORME, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Robert Debré, Paris, France

IPD SHARING:
Plan to Share IPD: No